CLINICAL TRIAL: NCT03265431
Title: Evaluation of PET/MR in Patients Selected for Ablation Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Marc D.Normandin, Ph.D, Associate Professor, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016P002123
Record Dates: First submitted 2017-08-25; First posted 2017-08-29 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Normal subjects without history of cardiac disease or arrhythmia
  Interventions: Drug: 18F-TPP
- Arrhythmia (Experimental): This cohort consist of patients with history of recurrent VT and scheduled for EAM-guided catheter ablation as part of their clinical treatment
  Interventions: Drug: 18F-TPP
- Treatment Failure (Experimental): A subset of the Arrhythmia cohort, this group will undergo a second imaging session. This subset corresponds to patients from the Arrhythmia cohort presenting with recurrent ventricular arrhythmia following initial EAM-guided catheter ablation and requiring repeated ablation. It is estimated that 30% of the Arrhythmia cohort patients will require repeat ablation based on rate of repeat ablation procedures at MGH. T
  Interventions: Drug: 18F-TPP

INTERVENTIONS:
Drug: 18F-TPP — Imaging with 18-F-TPP (18F-BFPET)
  Other Names: 18F-BFPET

SUMMARY:
This study is performed to assess if PET-MR imaging can improve treatment of patients with irregular heart rate and heart failure. Heart failure occurs when the heart muscle is too weak to do his work correctly. Irregular heart rate can be related to numerous diseases. One category of irregular heart rate is called ventricular arrhythmia. It is often seen in patients who have had a heart attack. This type of arrhythmia can be dangerous and can cause sudden death. To prevent these arrhythmias, doctors can perform procedures that burn the source of arrhythmia in the heart muscle. This is called ablation. Unfortunately, ablation does not fix the problem in 100% of patients and some will still have the arrhythmia requiring repeated procedure. The purpose of this study is to find new ways of guiding the doctors performing ablation, hoping to improve the success rate of the procedure.

ELIGIBILITY:
Healthy Volunteers

Inclusion Criteria:

* Subjects must be ≥21 and ≤80 years of age;
* Subjects must provide informed consent prior to study procedures;

Exclusion Criteria:

* Known structural heart disease (e.g. myocardial infarction);
* History of ventricular arrhythmia;
* Any contraindication to MRI and/or PET, including:
* Subjects with life vest;
* Subjects with implanted heart device (e.g. ICD, Pacemaker);
* Subjects with metallic fragment or foreign body;
* Subjects with other form of devices or prosthesis that are not MRI compatible, such as insulin pump, joint replacement, hearing aid, cochlear implant, permanent contraceptive devices, etc.;
* Claustrophobia;
* Relative or absolute contraindication to Dotarem contrast:
* history of renal disease including acute or chronic severe renal insufficiency (glomerular filtration rate <60 mL/min/1.73m2);
* a history of diabetes mellitus, systemic lupus, multiple myeloma, nephrogenic systemic fibrosis, and other co-morbidities;
* History of hypersensitive reactions to Dotarem and/or gadolinium contrast agent
* Any clinically significant acute or unstable physical or psychological disease, judged by the investigators based on medical history or screening physical examination, to be incompatible with the study;
* Any physical or psychological disease judged by the investigators to be incompatible with the study, based on medical history or screening physical examination
* Radiation exposure exceeds current Radiology Department guidelines (i.e. 50 mSv in the prior 12 months);
* Female subjects only: Positive serum and/or urine pregnancy test, or lactating, or possibility of pregnancy cannot be ruled out prior to dosing;
* Inability to provide written informed consent;

Arrhythmia Subjects:

Inclusion criteria

* Subjects must be ≥21 and ≤80 years of age;
* Subjects must provide informed consent prior to study procedures;
* History of scar-mediated ventricular arrhythmia scheduled for invasive EAM-guided catheter ablation for clinical care

Exclusion criteria

* Any contraindication to MRI and/or PET, including:
* Subjects with life vest;
* Subjects with implanted heart device (e.g. ICD, Pacemaker);
* Subjects with metallic fragment or foreign body;
* Subjects with other form of devices or prosthesis that are not MRI compatible, such as insulin pump, joint replacement, hearing aid, cochlear implant, permanent contraceptive devices, etc.;
* Claustrophobia;
* Relative or absolute contraindication to Dotarem contrast:
* history of renal disease including acute or chronic severe renal insufficiency (glomerular filtration rate <60 mL/min/1.73m2);
* history of diabetes mellitus, systemic lupus, multiple myeloma, nephrogenic systemic fibrosis, and other co-morbidities;
* History of hypersensitive reactions to Dotarem and/or gadolinium contrast agent;Any clinically significant acute or unstable physical or psychological disease, judged by the investigators based on medical history or screening physical examination, to be incompatible with the study;
* Any physical or psychological disease judged by the investigators to be incompatible with the study, based on medical history or screening physical examination
* Radiation exposure exceeds current Radiology Department guidelines (i.e. 50 mSv in the prior 12 months);
* Female subjects only: Positive serum and/or urine pregnancy test, or lactating, or possibility of pregnancy cannot be ruled out prior to dosing;
* Inability to provide written informed consent;

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
TPP imaging in Ventricular Arrhythmia | 5 years
  Establish imaging patterns allowing prediction of VT ablation failure

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pelletier-Galarneau M, Petibon Y, Ma C, Han P, Kim SJW, Detmer FJ, Yokell D, Guehl N, Normandin M, El Fakhri G, Alpert NM. In vivo quantitative mapping of human mitochondrial cardiac membrane potential: a feasibility study. Eur J Nucl Med Mol Imaging. 2021 Feb;48(2):414-420. doi: 10.1007/s00259-020-04878-9. Epub 2020 Jul 27. PMID 32719915